CLINICAL TRIAL: NCT05183542
Title: Predictive Performance of SPECT/CT Bone Scan Quantification Before Lumbar Arthrodesis
Brief Title: SPECT/CT Bone Scan Quantification Surgery
Acronym: PERQUAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Achraf BAHLOUL, MD, Central Hospital, Nancy, France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2021PI050
Record Dates: First submitted 2021-12-21; First posted 2022-01-10 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Pseudoarthrosis of Bone

STUDY DESIGN:
Intervention Model Description: Persons to be operated on for lumbar arthrodesis by the neurosurgery team of the Nancy CHRU and respecting the eligibility criteria (including neuropathic pain scale score < 4, see non-inclusion criteria), will be proposed to participate in the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Experimental): Patients with bone scan
  Interventions: Drug: Bone scan

INTERVENTIONS:
Drug: Bone scan — Persons to be operated on for lumbar arthrodesis by the neurosurgery team of the Nancy CHRU and respecting the eligibility criteria (including a score of neuropathique pain scale < 4, see non-inclusion criteria), will be proposed to participate in the study neuropathic pain If they give their oral agreement to the neurosurgeon, a request for a bone scan will be sent to the nuclear medicine department of the Nancy-Brabois Hospital. The patients will fill pain scales before and after surgery (ODI and NS)
  Other Names: Scales of pain

SUMMARY:
The hypothesis of our study is that SPECT/CT bone scan fixation quantified by SUVMAX on a CZT solid state camera preoperatively would identify good responders to lumbar arthrodesis surgery.

DETAILED DESCRIPTION:
Chronic low back pain is a public health problem and is the leading cause of work stoppage and the management of low back pain refractory to medical treatment involves surgical procedures such as arthrodesis, aimed at fusing several adjacent vertebrae.

The main gold standard tests for assessing the effectiveness of surgery are the Oswestry Disability Index (ODI), which takes into account the impact on quality of life and the numerical pain scale (EN). The ODI consists of 10 questions In order to compensate for the effect of analgesics on the ODI and EN scores, the response to both questionnaires should take into account the patient's symptomatology throughout the previous week.

A decrease in the score of these 2 scales by at least the value of the MCID (Minimal Clinically Important Difference) is necessary to conclude a good response to surgery . The MCID value is 10% (0-100% score) for the Oswestry Disability Index (ODI) and 19 points (0-100 point scale) for the Numerical Pain Scale (EN) respectively. Standard diagnostic investigations performed during the preoperative workup for arthrodesis, mainly include X-rays, CT and lumbar MRI but not bone scans. None of the current standard preoperative examinations can identify a group of people without improvement after surgery. semiconductor cameras, allow bone scans with CT recordings coupled to a CT scan (SPECT/CT) offering better performance compared to a conventional camera . If abnormalities are detected, the binding intensity of the radiopharmaceutical is not only assessed visually but can also be quantified by the Standardized Uptake Value (SUV).

To date, no preoperative examination that can predict the clinical evolution after lumbar arthrodesis has been reported apart from bone scintigraphy with visual assessment of fixation. Finding a threshold value for SUVmax to predict clinical outcome after surgery would potentially have an impact on the selection of "good responders" to lumbar spine arthrodesis, with other patients benefiting from medical treatment combined with rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Persons with back pain for at least 3 months (presumed to be due to degenerative disc disease or spondylolisthesis).
* Persons who have received full information about the organisation of the research and have signed the informed consent and :

  * Age ≥ 18 years, having read and understood the information document.
  * Affiliated to a social security scheme.
* Lumbar arthrodesis involving a maximum of 2 floors.
* Standardized lumbar arthrodesis surgery performed by one of the three senior neurosurgeons of the neurosurgery department of the Nancy CHRU, using similar surgical techniques.

Exclusion Criteria:

* Low back pain of neuropathic origin. The Neuropathic Pain Scale 4 questionnaire is used to diagnose neuropathic pain (score is ≥ 4/10)
* History of lumbar spine surgery
* Presence of other pathologies responsible for lumbar pain (multistage discopathies, ankylosing spondylitis, spondylodiscitis, rheumatoid arthritis, vertebral compression, vertebral metastasis, narrow lumbar canal, scoliosis, spondylolisthesis by isthmic lysis)
* Pregnant women or women of childbearing age without suitable contraception or nursing mothers.
* Unstable medical condition and/or inability to remain immobile in supine position during recordings.
* Known allergy to any component of the radiopharmaceutical (TECHNESCAN HDP).
* Person referred to in Articles L. 1121-5, L. 1121-7 and L1121-8 of the Public Health Code.
* Persons deprived of their liberty by a judicial or administrative decision, persons under psychiatric care by virtue of Articles L. 3212-1 and L. 3213-1.
* Persons of full age who are unable to express their opposition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-04-29 (Actual); Primary Completion 2025-11-29 (Estimated); Study Completion 2025-11-29 (Estimated)

PRIMARY OUTCOMES:
To determine if there is a correlation of SUV value and response to surgery with ODI | 24 months
  To determine whether SUVmax (Standard Uptake Value) measured at late time on bone scan, predicts a good response to lumbar arthrodesis surgery according to the Oswestry Disability Index (ODI) measured at 12 months after surgery

SECONDARY OUTCOMES:
To determine if there is a correlation of SUV value and response to surgery with NS | 24 months
  To determine whether SUVmax (Standard Uptake Value) measured at late time on bone scan, predicts a good response to lumbar arthrodesis surgery according to the numeric scale (NS) measured at 12 months after surgery
To determine if there is a correlation of SUV value at early time and response to surgery with ODI | 24 months
  To determine whether SUVmax measured at early time on bone scans predicts a good response to lumbar spine fusion surgery according to the Oswestry Disability Index (ODI) measured at 12 months after surgery.
To determine if there is a correlation of SUV value at early time and response to surgery with NS | 24 months
  To determine whether SUVmax measured at early time on bone scans predicts a good response to lumbar spine fusion surgery according to the Numeric Scale (NS) measured at 12 months after surgery.with Numeric Scale (NS)

CONTACTS AND LOCATIONS:
Overall Officials: El Mehdi SIAGHY, PhD, Study Director — CHRU Nancy
Locations (1):
- Nuclear Medicine Department, Vandœuvre-lès-Nancy, France